CLINICAL TRIAL: NCT02170220
Title: A Phase 1, Open-Label, Parallel-Group Study to Evaluate the Pharmacokinetics, Safety and Tolerability of a Single Oral Dose of 5 mg Vortioxetine in Subjects With Normal Hepatic Function or Severe Hepatic Impairment
Brief Title: Pharmacokinetics, Safety and Tolerability of Vortioxetine in Normal Hepatic Function or Severe Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LuAA21004_401; U1111-1155-8776 (Other: World Health Organization)
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Results first posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-12

CONDITIONS: Severe Hepatic Impairment
Keywords: Drug therapy
MeSH Terms: interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vortioxetine 5 mg: Normal Hepatic Function Cohort (Experimental): Vortioxetine 5 mg, tablets, orally, once, on Day 1, in participants with normal hepatic function.
  Interventions: Drug: Vortioxetine
- Vortioxetine 5 mg: Severe Hepatic Impairment Cohort (Experimental): Vortioxetine 5 mg, tablets, orally, once, on Day 1, in participants with severe hepatic impairment.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Vortioxetine tablets
  Other Names: Lu AA21004; BRINTELLIX

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of vortioxetine and its metabolites Lu AA34443 and Lu AA39835 following a single oral dose administration of vortioxetine 5 mg in participants with severe hepatic impairment compared to healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called vortioxetine. Vortioxetine is being tested to assess how it moves throughout the body in people with severe hepatic impairment compared to people with normal hepatic function. This study looked at lab results in people who took vortioxetine.

The study enrolled 12 participants. Participants were assigned to one of the two treatment groups based on their hepatic function (severe hepatic impairment vs. normal hepatic function). All participants in both groups will receive one vortioxetine 5-mg tablet.

This single-center trial was conducted in the United States. The overall time to participate in this study was up to 58 days. Participants made 2 visits to the clinic, including one 12-day period of confinement to the clinic, and were contacted by telephone 30 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

General:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is aged 18 to 75 years, inclusive, at the time of informed consent and first study medication dose.
4. Weighs at least 50 kg and has a body mass index (BMI) between 19 and 38 kg/m^2, inclusive at Screening.
5. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after last dose.
6. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study.
7. Has a resting pulse and heart rate (as read on electrocardiogram [ECG]) between 51 and 100 beats per minutes (bpm), inclusive. For healthy participants in good physical condition and aged 18 to 45 years, inclusive, the lower limit is 45 bpm.
8. Has a negative result at screening on the fecal occult blood screen.

   Healthy Participants (Normal Hepatic Function):
9. The participant, in opinion of the investigator, is in good health as determined by a prestudy physical examination, medical history, vital signs, ECG, and the results of blood biochemistry, hematology, and serology tests, and urinalysis.

   Participants with severe hepatic impairment:
10. Has been classified as having severe hepatic impairment as defined by the Child-Pugh classification system.
11. Has case record notes demonstrating stable biochemistry as judged by the investigator prior to Screening.
12. Has case record notes demonstrating physical signs consistent with a clinical diagnosis of liver impairment (eg, liver firmness to palpation, splenic enlargement, spider angiomas, palmar erythema, parotid hypertrophy, testicular atrophy, ascites, gynecomastia).
13. For participants with hepatic encephalopathy, the condition does not, in the investigator's opinion, interfere with the participant's ability to provide an appropriate informed consent. (Participants who have severe encephalopathy receive a score of 3 or 4. The score reflects the degree of encephalopathy off treatment. This will be documented in the source.)

Exclusion Criteria:

General:

1. Has received any investigational compound within 45 days prior to first dose of study medication.
2. Has received vortioxetine (Lu AA21004) in a previous clinical study or as a therapeutic agent.
3. Is an immediate family member, study site employee, or in a dependant relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has received or donated more than 400 mL of blood or blood products within the 45 days preceding the beginning of the study or planned to donate blood during the study.
5. Has a history of hypersensitivity or allergies to vortioxetine or related compounds with same mechanism of action including any associated excipients.
6. Has a medical history of, or presence of, gastric or duodenal ulceration, gastritis, recent head injury or any other trauma within 1 week of Screening, extensive ecchymoses, hemoptysis, gingival bleeding, hematemesis, repeated or significant nose bleeds, periorbital hematoma, retinal detachment, menorrhagia, hematuria, or melena.
7. Has had an acute, clinically significant illness within 30 days prior to the first dose of study medication.
8. Has a history of abdominal surgery (except laparoscopic cholecystectomy or uncomplicated appendectomy), thoracic, or nonperipheral vascular surgery within 6 months prior to the study medication.
9. Has a history of cancer, other than basal cell or Stage 1 squamous cell carcinoma of the skin that has not been in remission for at least 5 years prior to the first dose of study drug.
10. Has taken any medications, supplements or food products except for those allowed for hepatically impaired participants, or approved by Takeda on a case-by-case basis.
11. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 30 days after participating in this study; or intending to donate ova during such time period.
12. If male, the participant intends to donate sperm during the course of this study or for 30 days thereafter.
13. Has poor peripheral venous access.
14. Has a serum creatinine level greater than 1.5 mg/dL at Screening or Day -1 (Check-in).
15. Has active stage 3 or 4 encephalopathy.
16. Has a diastolic blood pressure >100 mm Hg or a systolic blood pressure >160 mm Hg (supine) at Screening or Day -1.
17. Has an orthostatic blood pressure ≥25 mm Hg (based on the difference between supine and standing [1 minute] systolic blood pressure) at Screening or Day 1.
18. Has a known history of human immunodeficiency virus infection.
19. Has a positive test result for hepatitis B surface antigen.
20. The participant's corrected QT interval (QTc, Bazett correction) is >450 millisecond (msec) for men and >470 msec for women at Screening or at Check-in as read on the printout of the ECG and evaluated by the investigator.
21. Has a history or clinical manifestations of significant illness such as renal insufficiency, hematologic, pulmonary, cardiovascular, gastrointestinal, neurological, rheumatologic, urologic, immunologic, infectious, skin and subcutaneous tissue disorders, or psychiatric or mood disorders (including any past suicide attempt). For hepatically impaired participants, previously known conditions associated with liver disease are not excluded.
22. Exercises extensively in his/her normal life, that is, marathon running, triathlons, physical sports at a contest level, etc.
23. Answers positive to any suicidal ideation and/or suicidal behavior questions during administration of the Columbia-Suicide Severity Rating Scale (C-SSRS) [7-9] at Screening.
24. Is unwilling or unable to comply with the protocol or scheduled appointments.
25. Is unable to understand verbal and/or written English or any other language for which a certified translation of the approved informed consent is available.
26. The participant, in the opinion of the investigator, is unlikely to comply with the clinical trial protocol or deemed unsuitable for any other reason.
27. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 2 alcoholic units per day) within 1 year prior to the Screening Visit (1 unit=250 mL of beer or 20 mL of spirits or 1 glass [118 mL] of wine). Participants with severe hepatic dysfunction who test positive on the urine drug screen due to prescription drug use will be allowed to participate if approved by the principal investigator and the sponsor's medical monitor.

    Healthy Participants (Normal Hepatic Function):
28. Has any clinically significant abnormal findings on the medical history, physical exam, ECG, or clinical laboratory tests that, in the opinion of the investigator, preclude study participation.
29. Has a hepatic and/or endocrine disorder.
30. Has a positive test result for antibody to hepatitis C virus.
31. Has an alanine transaminase or aspartate transaminase level of greater than 1.5 × upper limit of normal (ULN) at Screening or Day -1 (Check-in), active liver disease, active gall bladder disease, or jaundice.
32. Has a predisposition to easy bruising or bleeding, anemia, thrombocytopenia, or a known history, or history in a first-degree relative, of bleeding disorders (including Von Willebrand's disease or hemophilia A and B).
33. Has a positive test for fecal occult blood.

    Participants with severe hepatic impairment:
34. Has clinically significant laboratory abnormalities except for those parameters influenced by hepatic impairment.
35. Has any serious illness except for controlled hypertension or diabetes and those problems associated with the primary diagnosis of hepatic impairment or other diseases that are approved by the principal investigator and the sponsor's medical monitor.
36. Has a clinical exacerbation of liver disease (i.e, abdominal pain, nausea, vomiting, anorexia, or fever) within the 2-week period before the administration of study drug.
37. Has clinical demonstrable, massive, tense ascites.
38. Has evidence of acute viral hepatitis within 1 month prior to the administration of study medication.
39. Has evidence of hepatorenal syndrome.
40. Has a known history of bleeding disorders (including Von Willebrand's disease or hemophilia A and B).
41. Has active alcohol abuse or dependence as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- University of Miami, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 09 July 2014 (first participant signed the informed consent form) to 01 December 2014.
Pre-assignment Details: Participants with normal hepatic function and participants with severe hepatic impairment received a single dose of 5 mg vortioxetine.
Period: Overall Study
Arm/Group | Vortioxetine 5 mg: Normal Hepatic Function Cohort | Vortioxetine 5 mg: Severe Hepatic Impairment Cohort
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vortioxetine 5 mg: Normal Hepatic Function Cohort | Vortioxetine 5 mg: Severe Hepatic Impairment Cohort | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (2.58) | 54.8 (6.79) | 52.6 (5.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 5 | 10
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
Height [Mean (Standard Deviation); unit: cm] | 169.3 (10.31) | 165.7 (10.41) | 167.5 (10.06)
Weight [Mean (Standard Deviation); unit: kg] | 80.65 (13.261) | 82.17 (29.038) | 81.41 (21.537)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.02 (2.927) | 29.43 (7.554) | 28.73 (5.512)
Smoking Classification [Number; unit: participants]
  Never smoked | 5 | 3 | 8
  Current smoker | 1 | 1 | 2
  Ex-smoker | 0 | 2 | 2
Alcohol Classification [Number; unit: participants]
  Never drank | 5 | 3 | 8
  Current drinker | 1 | 3 | 4
  Ex-drinker | 0 | 0 | 0
Caffeine Consumption [Number; unit: participants]
  Yes | 3 | 3 | 6
  No | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Vortioxetine
Description: (AUC(0-tlqc) is a measure of total plasma exposure to the drug from time 0 to time of the last quantifiable concentration (AUC[0-tlqc]).
Time Frame: Predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, and 240 hours postdose
Population: Pharmacokinetic (PK) Analysis Set included all enrolled participants who received at least 1 dose of study drug with at least 1 measureable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Vortioxetine 5 mg: Normal Hepatic Function Cohort | Vortioxetine 5 mg: Severe Hepatic Impairment Cohort
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 166.955 (45.1656) | 188.663 (68.5380)

2. Primary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Vortioxetine Metabolite Lu AA34443
Description: as for outcome 1
Time Frame: Predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, and 240 hours postdose
Population: PK Analysis Set included all enrolled participants who received at least 1 dose of study drug with at least 1 measureable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Vortioxetine 5 mg: Normal Hepatic Function Cohort | Vortioxetine 5 mg: Severe Hepatic Impairment Cohort
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 88.614 (53.1478) | 71.942 (48.9356)

3. Primary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Vortioxetine Metabolite Lu AA39835
Description: as for outcome 1
Time Frame: Predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, and 240 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Vortioxetine 5 mg: Normal Hepatic Function Cohort | Vortioxetine 5 mg: Severe Hepatic Impairment Cohort
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 1.143 (1.2640) | 0.078 (0.1903)

4. Primary Outcome: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Vortioxetine
Description: AUC(0-inf) is a measure of total plasma exposure to the drug from time zero extrapolated to infinity.
Time Frame: Predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, and 240 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Vortioxetine 5 mg: Normal Hepatic Function Cohort | Vortioxetine 5 mg: Severe Hepatic Impairment Cohort
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 187.202 (52.8692) | 288.053 (148.7612)

5. Primary Outcome: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Vortioxetine Metabolite Lu AA34443
Description: AUC(0-inf) is a measure of total plasma exposure to the drug from time zero extrapolated to infinity.
Time Frame: Predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, and 240 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Vortioxetine 5 mg: Normal Hepatic Function Cohort | Vortioxetine 5 mg: Severe Hepatic Impairment Cohort
Number analyzed (Participants) | 5 | 5
ng*hr/mL | 122.899 (39.2417) | 124.708 (46.8665)

6. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Vortioxetine
Description: Maximum Observed Plasma Concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, and 240 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vortioxetine 5 mg: Normal Hepatic Function Cohort | Vortioxetine 5 mg: Severe Hepatic Impairment Cohort
Number analyzed (Participants) | 6 | 6
ng/mL | 2.078 (0.4675) | 1.670 (0.6135)

7. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Vortioxetine Metabolite Lu AA34443
Description: as for outcome 6
Time Frame: Predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, and 240 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vortioxetine 5 mg: Normal Hepatic Function Cohort | Vortioxetine 5 mg: Severe Hepatic Impairment Cohort
Number analyzed (Participants) | 6 | 6
ng/mL | 2.654 (1.6018) | 1.374 (0.7849)

8. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Vortioxetine Metabolite Lu AA39835
Description: as for outcome 6
Time Frame: Predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, and 240 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vortioxetine 5 mg: Normal Hepatic Function Cohort | Vortioxetine 5 mg: Severe Hepatic Impairment Cohort
Number analyzed (Participants) | 6 | 6
ng/mL | 0.029 (0.0324) | 0.008 (0.0190)

9. Primary Outcome: AUC(0-tlqc)u: Area Under the Unbound Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Vortioxetine
Description: AUC(0-tlqc)u is a measure of total unbound plasma exposure to the drug from time 0 to time of the last quantifiable concentration (AUC[0-tlqc]u).
Time Frame: Predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, and 240 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Vortioxetine 5 mg: Normal Hepatic Function Cohort | Vortioxetine 5 mg: Severe Hepatic Impairment Cohort
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 1.611 (0.4937) | 1.653 (0.6882)

10. Primary Outcome: AUC(0-inf)u: Area Under the Unbound Plasma Concentration-time Curve From Time 0 to Infinity for Vortioxetine
Description: AUC(0-inf)u is a measure of total unbound plasma exposure to the drug from time zero extrapolated to infinity.
Time Frame: Predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, and 240 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Vortioxetine 5 mg: Normal Hepatic Function Cohort | Vortioxetine 5 mg: Severe Hepatic Impairment Cohort
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 1.806 (0.5685) | 2.558 (1.5242)

11. Primary Outcome: Cmaxu: Maximum Observed Unbound Plasma Concentration for Vortioxetine
Description: Maximum Observed Unbound Plasma Concentration (Cmaxu) is the peak unbound plasma concentration of a drug after administration, obtained directly from the unbound plasma concentration-time curve.
Time Frame: Predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, and 240 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vortioxetine 5 mg: Normal Hepatic Function Cohort | Vortioxetine 5 mg: Severe Hepatic Impairment Cohort
Number analyzed (Participants) | 6 | 6
ng/mL | 0.020 (0.0056) | 0.014 (0.0053)

ADVERSE EVENTS:
Time Frame: The first dose of study drug to within 32 days
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Vortioxetine 5 mg: Normal Hepatic Function Cohort | Vortioxetine 5 mg: Severe Hepatic Impairment Cohort
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine 5 mg: Normal Hepatic Function Cohort (N=6) | Vortioxetine 5 mg: Severe Hepatic Impairment Cohort (N=6)
Vomiting (Gastrointestinal disorders) | 0 | 1
Blood potassium increased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be made without Sponsor's prior written approval. Any proposed publication or presentation will be submitted to Sponsor for review 60 days in advance of publication. Institution will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for an additional 60 days to preserve intellectual property.